CLINICAL TRIAL: NCT06725225
Title: Development of a Machine Learning-Based Risk Prediction Model and Stratified Management Strategies for Quality of Life in Lung Cancer Patients Undergoing Immunotherapy
Brief Title: Machine Learning for Predicting and Managing Quality of Life in Lung Cancer Immunotherapy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Zunyi Medical University (Other)
Collaborators: Ministry of Education of the People's Republic of China, Department of Humanities and Social Sciences (Unknown)
Responsible Party: Principal Investigator, Jian-Guo Zhou, MD, PhD, associate professor and associate chief physician, Second Affiliated Hospital of Zunyi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24YJCZH462
Record Dates: First submitted 2024-12-01; First posted 2024-12-10 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer Patients
Keywords: HRQOL; lung cancer; immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: A symptom cluster care intervention plan is being developed, and a research team is formed. Based on relevant literature and qualitative interviews, and guided by symptom management theory and the Knowledge-Attitude-Practice (KAP) behavior model, an initial draft of the care intervention plan is created and refined through expert consultation to finalize the plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The group with milder symptoms and better quality of life (Placebo Comparator): the group uses unsupervised machine learning to identify patients with severe symptoms and poor functionality who are receiving immunotherapy for non-small cell lung cancer, and implements a symptom cluster care intervention.
  Interventions: Behavioral: Conventional care intervention
- The group with more severe symptoms and poorer quality of life (Active Comparator)
  Interventions: Behavioral: Symptom cluster-based care intervention

INTERVENTIONS:
Behavioral: Symptom cluster-based care intervention — The patient symptoms were surveyed to develop a symptom cluster care intervention plan. The specific steps were as follows: a research team was established, relevant literature was reviewed, and qualitative interviews were conducted. Guided by symptom management theory and the Knowledge-Attitude-Practice (KAP) behavior model, a draft of the care intervention was created. This draft was then refined through expert consultation to finalize the intervention plan.
  Arms: The group with more severe symptoms and poorer quality of life
Behavioral: Conventional care intervention — Standard nursing intervention. This refers to routine clinical care without a specific care plan tailored to the patient's symptoms. For example, if a patient has symptoms, the nurse assists the patient in notifying the doctor but does not provide any special treatment themselves
  Arms: The group with milder symptoms and better quality of life

SUMMARY:
The goal of this study is to explore whether health-related quality of life (HRQoL) can be used as a predictive indicator for lung cancer patients and to implement clinical interventions. The study addresses two main objectives:

Analyzing HRQoL data of lung cancer patients undergoing immunotherapy using machine learning clustering methods to explore data patterns and build an HRQoL early warning model (already developed).

Validating this HRQoL early warning model in real-world settings by classifying patients with different HRQoL characteristics and assessing the clinical value of the model

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer incidence and mortality in China, and it holds the same position in the United States. Non-small cell lung cancer (NSCLC) is the most common histological type, accounting for approximately 85% of lung cancer cases. Treatment strategies based on pathology, molecular subtyping, and clinical staging include surgery, radiotherapy, chemotherapy, targeted therapy, and immunotherapy. In recent years, immunotherapy has been extensively researched and applied in lung cancer treatment. It works by blocking the binding of PD-L1 on tumor cells to PD-1 on T cells, thereby releasing the inhibition of T cell function and killing the tumor cells. Immunotherapy has become the standard treatment for advanced NSCLC without driver mutations, and it covers the entire spectrum of non-surgical locally advanced NSCLC consolidation therapy, perioperative neoadjuvant, and adjuvant therapy for early-stage NSCLC. However, not all patients benefit from immunotherapy, with only a small subset experiencing clinical benefit. Therefore, identifying resistance mechanisms, selecting populations that benefit from treatment, and overcoming therapy resistance are complex and challenging clinical issues that require collaboration among basic, translational, and clinical oncology research teams.

In 1993, the World Health Organization (WHO) introduced the concept of Quality of Life (QoL), which refers to an individual's perception of their position in life within their cultural and value system, relating to their goals, expectations, standards, and concerns. Few studies focus on cancer patients' QoL, particularly those using patient-reported outcomes (PRO) as a primary endpoint. Most clinical trials for cancer drugs use PROs as secondary or exploratory endpoints. There is limited research that considers PROs as the primary endpoint. Therefore, it is essential to further investigate the relationship between cancer patients' health-related quality of life and prognosis, as well as its relevance to immunotherapy. This would facilitate better early identification of immune-related adverse events and systematic management, improving treatment adherence, QoL, and ensuring optimal treatment outcomes.

This project aims to develop a risk warning model for health-related quality of life in lung cancer patients receiving immunotherapy based on machine learning. By using cluster analysis, the study will clean, validate, and analyze the health-related quality of life data from the QLQ-C30 and QLQ-LC13 questionnaires from clinical trials available on the Vivli Global Clinical Research Data Sharing and Analysis Platform. The goal is to identify the distribution characteristics of these data and explore whether patient-reported outcomes can predict the efficacy of immunotherapy, thus serving as biomarkers to identify potential beneficiaries of immunotherapy. Furthermore, based on a risk warning and stratified management approach, the project aims to design appropriate symptom intervention strategies for different PRO types in immunotherapy patients, ultimately helping healthcare providers better understand the symptom burden that lung cancer patients may experience during immunotherapy and offering practical guidance for symptom management.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed with lung cancer
2. Age over 18 years
3. Currently receiving immunotherapy for lung cancer
4. Good verbal communication ability
5. Informed consent signed by the patient or family member

Exclusion Criteria:

1. Cognitive impairment or mental illness
2. Other severe diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ C30 | Two weeks after the intervention
  The EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30) is a tool used to assess the quality of life in cancer patients. It consists of 30 items covering functioning, symptoms, and overall health status. Scores for each item range from 0 to 4 or 0 to 7 (depending on the item type), with overall scores typically ranging from 0 to 100. Higher scores indicate better quality of life with fewer symptoms and better functioning, while lower scores reflect worse quality of life with more severe symptoms and poorer functioning.
EORTC QLQ LC-13 | Two weeks after the intervention
  The EORTC QLQ LC-13 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer Module 13) is a questionnaire used to assess the quality of life of lung cancer patients. It includes 13 items, with scores ranging from 0 to 4, and the total score ranges from 0 to 52. A higher score indicates more severe symptoms and poorer quality of life, while a lower score indicates better quality of life. The EORTC QLQ LC-13 is often used in conjunction with the EORTC QLQ-C30 scale, as they complement each other and provide a comprehensive assessment of the quality of life in lung cancer patients.

SECONDARY OUTCOMES:
ORR (Objective Response Rate) | Two weeks after the intervention
  ORR refers to the proportion of patients who achieve either a complete response (CR) or partial response (PR) during treatment. This endpoint reflects the effectiveness of the treatment in controlling the tumor. It is typically assessed through imaging techniques (e.g., CT, MRI) and scored based on RECIST (Response Evaluation Criteria in Solid Tumors) or similar criteria. ORR is a common efficacy endpoint in cancer clinical trials.
PFS (Progression-Free Survival) | Two weeks after the intervention
  PFS refers to the length of time from the start of treatment until the tumor progresses or the patient dies, typically assessed through imaging or clinical evaluation. This endpoint reflects the effectiveness of the treatment in delaying disease progression. PFS is particularly useful in evaluating the clinical efficacy of new drugs or therapies. An extension of PFS is usually considered a sign of effective treatment.

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- Available data/document: Individual Participant Data Set — https://vivli.org